CLINICAL TRIAL: NCT07043907
Title: A Single-center, Single-arm Exploratory Clinical Trial on the Safety and Efficacy of PANK-003 Cell Injection Combined With Standard Adjuvant Chemotherapy After Surgery in Patients With Stage IIIA Non-Small Cell Lung Cancer
Brief Title: PANK-003 Cell Injection Combined With Standard Adjuvant Chemotherapy After Surgery in Patients With Stage IIIA NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Celconta Life Science Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ETHICS COMMITTEE OPIN-038
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy (Experimental)
  Interventions: Drug: PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy

INTERVENTIONS:
Drug: PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy — PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy

SUMMARY:
A Single-center, Single-arm Clinical Trial on the Safety and Efficacy of PANK-003 Cell Injection Combined with Standard Adjuvant Chemotherapy After Surgery in Patients with Stage IIIA Non-Small Cell Lung Cancer

DETAILED DESCRIPTION:
This study is a single-center, single-arm, open-label, single-dose administration dose-finding study, which aims to evaluate the safety and efficacy characteristics of PANK-003 Cell Injection Combined with Standard Adjuvant Chemotherapy After Surgery in Patients with Stage IIIA Non-Small Cell Lung Cancer.

The study includes a screening period, a treatment period, and an observation and follow-up period.

The main objectives :

To evaluate the safety and efficacy of multiple injections of PANK-003 cell injection combined with standard postoperative adjuvant chemotherapy in the treatment of patients with Stage IIIA Non-Small Cell Lung Cancer.

Primary Endpoints： Safety Endpoints: Incidence and severity of investigator-assessed adverse events (AEs), and clinically significant abnormal laboratory findings.

Efficacy Endpoint: 1-year DFS% assessed by the Independent Radiology Review Committee according to RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical trial; fully understand and be informed about this study and sign the informed consent form;
2. At the time of screening, the age should be between 18 and 75 years old (inclusive), regardless of gender;
3. Patients with histologically confirmed stage IIIA NSCLC (T4N0M0, T3-4N1M0, T1a-2bN2M0) who underwent R0 resection and received postoperative adjuvant chemotherapy (Exclusion of EGFR sensitizing mutations and ALK fusion); and who received the first dose of PANK-003 cell injection combined with postoperative adjuvant chemotherapy within 8 weeks after radical surgery.;
4. At the time of enrollment, the expected survival time is more than 6 Months;
5. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0 or 1;
6. At the time of screening, the laboratory tests should meet the following requirements:

   * White blood cell count ≥ 3.0×10⁹/L;
   * Neutrophil count ≥ 1.5×10⁹/L;
   * Lymphocyte count ≥ 0.5×10⁹/L;
   * Hemoglobin ≥ 90 g/L;
   * Platelets ≥ 75×10⁹/L;
   * Serum total bilirubin ≤ 2.0 × ULN (Upper Limit of Normal); for patients with a history/suspected Gilbert's syndrome, total bilirubin (TBIL) must be ≤ 3 × ULN.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN;
   * Creatinine < 1.5×ULN and endogenous creatinine clearance rate ≥ 50 mL/minute (Cockcroft-Gault method for calculating creatinine clearance rate: For men, creatinine clearance rate = [(140 - age) × body weight (kg)] / [0.818 × creatinine (μmol/L)]; For women, creatinine clearance rate = [(140 - age) × body weight (kg) × 0.85] / [0.818 × creatinine (μmol/L)]).
7. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and be willing to use medically recognized highly effective contraception during the study and for at least 1 year after the last study treatment; male subjects with partners of childbearing potential must have undergone surgical sterilization or agree to use effective contraception during the study and for at least 1 year after the last study treatment;
8. Investigator-confirmed eligibility for study enrollment.

Exclusion Criteria:

1. NSCLC patients who have received neoadjuvant therapy;
2. Pregnant or lactating women;
3. History of other malignancies, except:

   * Cured non-melanoma skin cancer
   * Carcinoma in situ of the cervix
   * Localized prostate cancer
   * Superficial bladder cancer
   * Other malignancies with disease-free survival >5 years;
4. Positive virology serology meeting any of:

   * HBsAg(+) and/or HBeAg(+) with HBe-Ab(+) and/or HBc-Ab(+) and HBV-DNA > lower limit of quantification
   * HCV-Ab(+)
   * TP-Ab(+)
   * HIV-Ab(+);
5. Received investigational drugs or other cell-based immunotherapy within 28 days before screening;
6. Administration of live/attenuated vaccines within 4 weeks prior to NK cell infusion;
7. Medical conditions requiring systemic corticosteroid therapy or other immunosuppressive drug treatments during the study period as determined by the investigator;
8. Hypersensitivity to:

   * Any component of NK cell products (including serum albumin)
   * Common emergency medications or anesthetics;
9. Unstable cardiovascular diseases within 180 days pre-screening, including:

   * Unstable angina
   * Myocardial infarction
   * Heart failure (NYHA class ≥III)
   * Severe arrhythmia requiring medication
   * Cardiac angioplasty, coronary stenting, or CABG;
10. Any condition that may compromise protocol compliance or patient safety as determined by the investigator:

    * Poorly controlled diabetes
    * Uncontrolled infections
    * Central nervous system disorders
    * Bleeding/thrombotic diathesis
    * Poor compliance
    * Substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-07-08 (Estimated); Primary Completion 2028-07-08 (Estimated); Study Completion 2029-06-18 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | 3 months
  Incidence, severity and clinically significant abnormal laboratory findings of treatment related AEs.
Disease Free Surviva Percentage（DFS%） | 1 year
  Disease Free Survival (DFS): The time from the first infusion day of PANK - 003 cell injection in subjects to the recurrence of the tumor (including local recurrence, regional recurrence, or distant metastasis) or death due to any cause.
  Disease Free Surviva Percentage（DFS%）: It refers to the proportion of subjects who have not experienced tumor recurrence or death at a specific follow-up time point, typically expressed as a percentage. Its core lies in using survival analysis methods, combined with the follow-up data of subjects, to estimate the disease-free survival probabilities at different time points.

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | 1 year
  Disease Free Survival (DFS): The time from the first infusion day of PANK - 003 cell injection in subjects to the recurrence of the tumor (including local recurrence, regional recurrence, or distant metastasis) or death due to any cause.
Overall Survival (OS) | 1 year
  Overall Survival (OS):The time from the date of first administration of PANK-003 cell injection to deathfrom any cause.
Tumor Recurrence Rate (TRR) | 1 year
  Tumor Recurrence Rate (TRR): The proportion of subjects who experience tumor recurrence from the first infusion day of PANK-003 to the end of follow-up.

IPD SHARING:
Plan to Share IPD: No